CLINICAL TRIAL: NCT04334486
Title: The Effects of Video Game Warm-up on EyeSi Surgical Simulator Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-0110
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: High Fidelity Simulation Training
Keywords: training effect; bimanual dexterity; surgical skills; ophthalmology

STUDY DESIGN:
Intervention Model Description: Non-blinded parallel examination of training or non-training effect of video game participation prior to Eyesi surgical simulator evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Game Trained (Experimental): Subjects will participate in video gaming for 10 minutes prior to Eyesi simulator test of surgical skills.
  Interventions: Other: Super Smash Brothers Melee (Gamecube)
- No Video Game Training (No Intervention): No video gaming will occur for warm up to Eyesi simulator test of surgical skills

INTERVENTIONS:
Other: Super Smash Brothers Melee (Gamecube) — 10 minutes of participation in Super Smash Brothers Melee prior to Eyesi Surgical Simulator evaluation of skills.
  Arms: Video Game Trained

SUMMARY:
This study will examine the history of video game use an activities of manual dexterity with the scored skills used in the Eyesi surgical simulator. Subjects will be asked to participate in video games or no video games prior to testing skills in Eyesi to examine training effects of video game participation and changes in manual dexterity.

DETAILED DESCRIPTION:
A popular crossover fighting video game released in 2001 for the Nintendo Gamecube that emphasizes reflexes and dexterity to perform specific maneuvers will be used in this study as a potential dexterity trainer.

The Eyesi is a training device utilized in many ophthalmology residency training programs to improve intraocular operative skills. The EyeSi is a validated training tool that uses high-end virtual reality that can be equipped with instrumentation for cataract or vitreoretinal surgery. The device itself consists of eyepieces that replicate a surgical scope, a mannequin head where handpiece probes can be inserted and position tracked to virtually recreate a surgical environment. The simulator also has a monitor that can be used to see the surgical simulator environment. As part of the software, numerous training tasks and exercises are available programmed into the device. These exercises utilize numerous metrics such as distance traveled, tissue treatment, efficiency, instrument handing, and others to provide the user with a raw score out of 100 for each task.

Subjects will then be asked to complete a manual dexterity questionnaire including history of video game use as well as tasks demonstrating manual dexterity ability such as the ability to play a musical instrument. Participants will then be randomized to the intervention group or the control group.

The intervention group will be asked to play 10 minutes of the Gamecube game "Super Smash Brothers Melee" as their "warm-up" prior to completing the EyeSi surgical tasks of navigation, forceps, and bimanual with their scores collected and averaged across all tasks.

The control group will complete the EyeSi surgical tasks of navigation, forceps, and bimanual with their scores collected and averaged, but will not perform a "warm-up" task.

Planned statistical analysis will include an average of total scores across navigation, forceps, and bimanual tasks. Chi square analysis will then be utilized to determine any statistical significance between intervention and control groups. Simulator scores will also be associated with questionnaire responses and simple linear regression will be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* UTMB Medical student volunteers who respond to email invitation to participate
* 18-40 years of age inclusive

Exclusion Criteria:

* Prior experience with EyeSi surgical simulator
* Not a UTMB Medical Student
* Not between 18-40 years of age inclusive

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Video Game training effect on Eyesi Surgical Simulator Scores | 30 minutes
  Planned statistical analysis will include an average of total scores across navigation, forceps, and bimanual tasks. Chi square analysis will then be utilized to determine any statistical significance between intervention and control groups.

SECONDARY OUTCOMES:
Training effect of manual dexterity activities on Eyesi Surgical Simulator Scores as reported in questionnaire. | 30 minutes
  Subjects will then be asked to complete a manual dexterity questionnaire including history of video game use as well as tasks demonstrating manual dexterity ability such as the ability to play a musical instrument. Simulator scores will be associated with questionnaire responses and simple linear regression will be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Praveena Gupta, M.D., Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Ophthalmology Clinical Research Center, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data will be assigned a unique participant identification number and no personal information will be collected as part of the data set. Information from the questionnaire and study tasks will be associated with your subject identification number not any personal identifiers. Your participation or lack of participation will not be made known to any individuals outside of the study personnel with which you interface and will also be unavailable to any faculty within the UTMB Ophthalmology program to ensure that there is no risk in participation affecting future departmental relationships, evaluations or considerations.

REFERENCES:
- [Background] Crochet P, Aggarwal R, Dubb SS, Ziprin P, Rajaretnam N, Grantcharov T, Ericsson KA, Darzi A. Deliberate practice on a virtual reality laparoscopic simulator enhances the quality of surgical technical skills. Ann Surg. 2011 Jun;253(6):1216-22. doi: 10.1097/SLA.0b013e3182197016. PMID 21516035
- [Background] McCannel CA, Reed DC, Goldman DR. Ophthalmic surgery simulator training improves resident performance of capsulorhexis in the operating room. Ophthalmology. 2013 Dec;120(12):2456-2461. doi: 10.1016/j.ophtha.2013.05.003. Epub 2013 Jun 21. PMID 23796766
- [Background] Pokroy R, Du E, Alzaga A, Khodadadeh S, Steen D, Bachynski B, Edwards P. Impact of simulator training on resident cataract surgery. Graefes Arch Clin Exp Ophthalmol. 2013 Mar;251(3):777-81. doi: 10.1007/s00417-012-2160-z. Epub 2012 Sep 25. PMID 23007233
- [Background] Seymour NE, Gallagher AG, Roman SA, O'Brien MK, Bansal VK, Andersen DK, Satava RM. Virtual reality training improves operating room performance: results of a randomized, double-blinded study. Ann Surg. 2002 Oct;236(4):458-63; discussion 463-4. doi: 10.1097/00000658-200210000-00008. PMID 12368674
- [Background] Thomsen ASS, Kiilgaard JF, Kjaerbo H, la Cour M, Konge L. Simulation-based certification for cataract surgery. Acta Ophthalmol. 2015 Aug;93(5):416-421. doi: 10.1111/aos.12691. Epub 2015 Feb 26. PMID 25722080
- [Background] Bergqvist J, Person A, Vestergaard A, Grauslund J. Establishment of a validated training programme on the Eyesi cataract simulator. A prospective randomized study. Acta Ophthalmol. 2014 Nov;92(7):629-34. doi: 10.1111/aos.12383. Epub 2014 Mar 11. PMID 24612448
- [Background] Solverson DJ, Mazzoli RA, Raymond WR, Nelson ML, Hansen EA, Torres MF, Bhandari A, Hartranft CD. Virtual reality simulation in acquiring and differentiating basic ophthalmic microsurgical skills. Simul Healthc. 2009 Summer;4(2):98-103. doi: 10.1097/SIH.0b013e318195419e. PMID 19444047
- [Background] Thomsen AS, Bach-Holm D, Kjaerbo H, Hojgaard-Olsen K, Subhi Y, Saleh GM, Park YS, la Cour M, Konge L. Operating Room Performance Improves after Proficiency-Based Virtual Reality Cataract Surgery Training. Ophthalmology. 2017 Apr;124(4):524-531. doi: 10.1016/j.ophtha.2016.11.015. Epub 2016 Dec 22. PMID 28017423
- [Background] Daly MK, Gonzalez E, Siracuse-Lee D, Legutko PA. Efficacy of surgical simulator training versus traditional wet-lab training on operating room performance of ophthalmology residents during the capsulorhexis in cataract surgery. J Cataract Refract Surg. 2013 Nov;39(11):1734-41. doi: 10.1016/j.jcrs.2013.05.044. PMID 24160383
- [Background] Adams BJ, Margaron F, Kaplan BJ. Comparing video games and laparoscopic simulators in the development of laparoscopic skills in surgical residents. J Surg Educ. 2012 Nov-Dec;69(6):714-7. doi: 10.1016/j.jsurg.2012.06.006. PMID 23111035
- [Background] Middleton KK, Hamilton T, Tsai PC, Middleton DB, Falcone JL, Hamad G. Improved nondominant hand performance on a laparoscopic virtual reality simulator after playing the Nintendo Wii. Surg Endosc. 2013 Nov;27(11):4224-31. doi: 10.1007/s00464-013-3027-z. Epub 2013 Jun 13. PMID 23760943